CLINICAL TRIAL: NCT04297878
Title: The BLIS Study: a Feasibility Study Assessing Compliance, Acceptability and Colonisation With Different Dosing Regimens of the Probiotic Supplement Streptococcus Salivarius K12 (Bactoblis®) in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 52107.P
Record Dates: First submitted 2020-02-28; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Sore Throat; Tonsillitis; Pharyngitis
MeSH Terms: conditions — Pharyngitis; Tonsillitis

STUDY DESIGN:
Intervention Model Description: Two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Taking two SsK12 lozenges at night on days 1, 7 and 14.
  Interventions: Dietary Supplement: probiotic supplement Streptococcus salivarius K12 (Bactoblis®)
- Group B (Active Comparator): One SsK12 daily at night for 14 days.
  Interventions: Dietary Supplement: probiotic supplement Streptococcus salivarius K12 (Bactoblis®)

INTERVENTIONS:
Dietary Supplement: probiotic supplement Streptococcus salivarius K12 (Bactoblis®) — Probiotic food supplement

SUMMARY:
Short title The BLIS study

Full title A feasibility study assessing compliance, acceptability and colonisation with different dosing regimens of the probiotic supplement Streptococcus salivarius K12 (Bactoblis®) in adults

Population 50 human adults with or without a history of significant sore throat in the past 12 months. We primarily aim to recruit participants with a history of sore throat, however we will also recruit healthy individuals if we are struggling to meet our recruitment target.

Interventions

Two groups will receive two different dosing regimens of Ssk12 probiotic oral lozenges:

* Group A: two SsK12 lozenges at night on days 1, 7 and 14.
* Group B: one SsK12 daily at night for 14 days. Throat swabs will be taken at baseline, and days 2, 7, 14, 21, 35

Objectives

1. To evaluate the prevalence of colonisation with SsK12 (as determined by real-time Polymerase Chain Reaction [PCR] and culture of participant-take whole-mouth swabs at pre-determined time points during the study)
2. To evaluate the acceptability of the two dosing regimens (as measured by participant-completed questionnaires)
3. To evaluate participants compliance with the two dosing regimens (as reported by participants during completion of the questionnaires)

Rationale SsK12 probiotic supplements are recognised as safe food ingredients, and there is preliminary evidence to support their use as prophylactic therapy to prevent episodes of pharyngo-tonsillitis. Existing clinical trials have all given SsK12 once daily over a period of months. It remains unclear whether a once-daily dosing regimen is needed in order to establish and maintain colonisation.

Study design This is a prospective study for which we will recruit healthy adult participants with and without a history of sore throat/ pharyngo-tonsillitis. We will evaluate [1] the acceptability and feasibility of two different dosing regimens of SsK12 supplements (taken as oral dissolvable lozenges), and [2] compare the prevalence of colonisation with SsK12 at various time points in order to determine how long colonisation is maintained following a loading dose. A baseline whole-mouth swab will be taken, and participants will be randomly assigned (in a 1:1 ratio) to one of two groups ('A' or 'B'). Group A will take two SsK12 lozenges at night on days 1, 7 and 14. Group B will take SsK12 at night for 14 days. Participants will be provided with instruction on how to perform a self-taken whole-mouth swab, and asked to take swabs on days 2, 7, 14, 21, and 35, and return these to the study team by post. They will also be asked to complete two short online questionnaires (on day 14 and day 35) about their compliance with the probiotic, as well as their views on the dosing regimen and other aspects of the study. Maintenance of colonisation will be assessed using analysis of the returned throat swabs. No follow-up will be undertaken after day 35.

Sample size Total = 50 (25 in group A, and 25 in group B)

Setting

1. NIHR Clinical Research Facility, Southampton General Hospital
2. Cowley Road Medical Practice, Oxford

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Fully conversant in the English language
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Willing to take SsK12 and return throat swabs according to the study protocol
* We primarily aim to recruit participants with a history of sore throat, however we will also recruit healthy individuals with no history of sore throat if we are struggling to meet our recruitment target of 50. We are defining a 'history' of sore throat as two or more episodes of significant (as judged by the participant) sore throat/pharyngo-tonsillitis episodes in the past 12 months. However, if we are struggling to recruit, a decision may be made by the chief investigator to alter this definition to one or more episodes in the last 12 months, after consultation with the study team.

Exclusion Criteria:

* Involvement in a study involving the receipt of an investigational medical product within 30 days prior to, or during, the study period.
* Active symptoms of sore throat or other infection at the time of recruitment
* Presence of a chronic disease/condition (such as those affecting the oropharynx) which, in the view of the investigator, might impact on colonisation, impede analysis of the study results, put the participant at increased risk, or impact on the ability of the participant to follow the study procedures
* Participant unable to give informed consent
* Any confirmed or suspected immunosuppressive or immunodeficient state, or use of immunosuppressant medication (including oral steroids) within the last 30 days
* History of allergic disease or reactions likely to be exacerbated by any of the study treatment
* Current smokers (including e-cigarettes/vaping)
* Any other clinically significant (as determined by the investigator) abnormality on clinical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-05 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of colonisation with SsK12 | During study involvement (days 1-35)
  To evaluate the prevalence of colonisation with SsK12 (as determined by real-time Polymerase Chain Reaction [PCR] and culture of participant-take whole-mouth swabs at pre-determined time points during the study)
Acceptability of dosing regimens | During study involvement (days 1-35)
  To evaluate the acceptability of the two dosing regimens as measured by participant questionnaires completed on day 14 and day 35 (which include questions on a 1-5 Likert scale, as well as an opportunity to write open comments),
Compliance with dosing regimens | During study involvement (days 1-35)
  To evaluate participants compliance with the two dosing regimens. This will be self-reported by participants as part of the questionnaires completed on day 14 and day 35.

IPD SHARING:
Plan to Share IPD: No